CLINICAL TRIAL: NCT03850626
Title: Validierung Des cSMS in Patienten Mit Allergischer Rhinokonjunktivitis (Baum- Und Gräserpollen, Hausstaubmilben). - Eine NIS Bei Patienten, Die Depigoid® Als Spezifische Immuntherapie Erhalten
Brief Title: Validation of Combined Symptom Medication Score (cSMS) in Allergic Patients
Status: Completed | Type: Observational
Sponsor: Leti Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: cSMS-2018
Record Dates: First submitted 2019-02-18; First posted 2019-02-22 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Allergic Rhinoconjunctivitis; Allergic Asthma
Keywords: Allergy; Rhinoconjuctivitis; Combined Symptom and Medication Score; Allergic Asthma; Pollen; Mites
MeSH Terms: conditions — Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immunotherapy Trees: Patients allergic to tree pollen
  Interventions: Biological: Immunotherapy
- Immunotherapy Grass: Patients allergic to grass pollen
  Interventions: Biological: Immunotherapy
- Immunotherapy Mites: Patients allergic to HDM
  Interventions: Biological: Immunotherapy

INTERVENTIONS:
Biological: Immunotherapy — subcutaneous injection

SUMMARY:
The CSMS was defined by the European Academy of Allergy and Immunology Taskforce as a standardised tool to assess clinical effects of allergen-specific immunotherapy (AIT). The aim of this study is to validate the CSMS as a tool to assess the clinical effects of Depigoid AIT, so that the CSMS can be used in future studies as a primary endpoint as well as a comparative parameter.

DETAILED DESCRIPTION:
Approximately 20% of the general public suffer from seasonal or perennial allergic rhinoconjunctivitis. The only available curative therapy is AIT. The effectiveness of AIT was demonstrated in numerous randomized clinical trials but comparability is difficult because of different primary and secondary endpoints.

To validate the CSMS, adolescent (≥ 12 years) and adult patients will be observed who are allergic to house dust mites (HDM), tree or grass pollen and who were treated with Depigoid. Depigoid is a registered (for tree and grass pollen) respective authorized (for HDM) suspension for injection for the treatment of immediate type allergic diseases. Depigoid contains depigmented and chemically modified allergen extracts, so called allergoids, derived from grass pollen, tree pollen or HDM.

Allergy symptoms will be documented over a time period of two years: Either for two consecutive allergy seasons (for tree and grass pollen allergic patients) or for two consecutive exposure periods (September-December) for HDM allergic patients. The symptoms (4 nasal and 2 ocular symptoms) and allergy medication intake will be documented on a daily basis either using the CSMS questionnaire or the especially developed electronic CSMS+ diary application.

Already validated and established questionnaires will be used to validate the CSMS with regard to Quality of Life (QoL) and symptom control: the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), Adolescent RQLQ (AdolRQLQ, for patients aged 12-17 years), Asthma Quality of Life Questionnaire (AQLQ) and AQLQ for patients aged 12 years and older (AQLQ+12), the Asthma Control Test (ACT), Rhinitis Control Assessment Test (RCAT) and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

- Indication of an allergen-specific immunotherapy with Depigoid

Exclusion Criteria:

- exclusion criteria according to the SmPC

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adults and adolescents suffering from allergic diseases (rhinitis, rhinoconjunctivitis, with or without concomitant asthma)
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
cSMS | after up to 60 days during allergen exposure period (=pollen season resp. allergen season) in 2 consecutive years
  Combined Symptom and Medication Score

CONTACTS AND LOCATIONS:
Overall Officials: Angelika Sager, Dr.med., Study Director — Medical Department
Locations (1):
- Dr. med Andrea Kienle-Gogolok, Bad Schönborn, Germany

IPD SHARING:
Plan to Share IPD: No